CLINICAL TRIAL: NCT06760585
Title: Prognostic Factors Associated With Failure of Total Elbow Replacement: a Protocol for Analysis of National Joint Registry Data
Brief Title: Prognostic Factors Associated With Failure of Total Elbow Replacement
Status: Not yet recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: The National Joint Registry (Unknown); The Royal College of Surgeons of England (Other); John Charnley Trust (Unknown); University of Bristol (Other)
Responsible Party: Principal Investigator, Zaid Hamoodi, National Joint Registry research fellow and PhD Student, University of Manchester
Other Study IDs: 7271373
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Total Elbow Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to evaluate potential prognostic factors for TER failure . The National Joint Registry (NJR) currently contains the largest elbow registry dataset in the world, which has been shown to have high completeness and accuracy. In order to incorporate additional potential prognostic factors not captured in the NJR, this study will combine the NJR elbow dataset with the NHS England Hospital Episode Statistics-Admitted Patient Care (HES-APC) data. Understanding prognostic factors is a crucial step for informing the development of strategies aimed at minimising the risk of failure and the necessity for additional surgery, which poses a burden on patients and society.

ELIGIBILITY:
Inclusion Criteria:

All patients aged 16 to 100 years old with a primary TER on the National Joint Registry (NJR) elbow dataset from the start of data collection on the 1st of April 2012 to the 31st of December 2023 will be included.

Exclusion Criteria:

Patients are excluded if they did not consent for their data to be used for research purposes, if it is impossible to trace them after surgery, if their ID numbers are invalid, or if the surgery was not performed in England.

Unconfirmed procedures and procedures with inconsistent operative patterns (i.e. a sequence of operations where the primary operation is not the first operation in the sequence or where there are multiple primary operations recorded for the same joint) will be excluded from the analyses.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with a primary total elbow replacement in England on the National Joint Registry (NJR)
Sampling Method: Non-Probability Sample
Enrollment: 4073 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
The hazard of failure of total elbow replacement | 11 years
  Indicated by the need for revision surgery recorded on the NJR. The NJR's definition of "revision surgery" will be used, which encompasses any operation involving the addition, removal, or modification of one or more components in a joint replacement. This includes debridement, antibiotics, and implant retention (DAIR) with modular exchange procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Epidemiology Versus Arthritis, Centre for Musculoskeletal Research, University of Manchester, Manchester Academic Health Science Centre, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The National Joint Registry (NJR) elbow data can be requested for research purposes through an application to the NJR research committee. Researchers do not have the rights to share the data directly

REFERENCES:
- [Derived] Hamoodi Z, Sayers A, Whitehouse MR, Kearsley-Fleet L, Sergeant JC, Watts AC. Prognostic factors associated with failure of total elbow replacement: a protocol for analysis of National Joint Registry data in England. BMJ Open. 2025 Jul 1;15(7):e098729. doi: 10.1136/bmjopen-2025-098729. PMID 40592743